CLINICAL TRIAL: NCT04356742
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Dapagliflozin When Added to Ongoing Metformin and Evogliptin Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Efficacy and Safety of Dapagliflozin When Added to Ongoing Metformin and Evogliptin Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA1229_DMTD2_III
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10mg + Evogliptin 5mg + Metformin (Experimental)
  Interventions: Drug: Dapagliflozin 10mg; Drug: Evogliptin 5mg; Drug: Metformin≥1000mg
- Dapagliflozin Placebo + Evogliptin 5mg + Metformin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Evogliptin 5mg; Drug: Metformin≥1000mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10mg, orally, once daily, up to 24weeks
  Other Names: Forxiga
  Arms: Dapagliflozin 10mg + Evogliptin 5mg + Metformin
Drug: Placebo — Dapagliflozin Placebo, orally, once daily, up to 24weeks
  Arms: Dapagliflozin Placebo + Evogliptin 5mg + Metformin
Drug: Evogliptin 5mg — Evogliptin 5mg, orally, once daily for background therapy
  Other Names: Suganon
Drug: Metformin≥1000mg — Metformin≥1000mg, orally, daily for background therapy

SUMMARY:
This study evaluates the addition of dapagliflozin in the treatment of type 2 diabetes with metformin and evogliptin combination therapy. Half of subjects will receive dapagliflozin, metformin and evogliptin, while the other half will receive placebo, metformin and evogliptin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type II diabetes mellitus aged 19 years or older
2. Patients who had taken metformin(≥1000mg/day) and DPP(dipeptidyl peptidase)-4 inhibitor combination therapy(or complex is allowed) at the same dose for at least 8 weeks prior to the screening visit
3. Patients with fasting plasma glucose≤250mg/dL at the screening visit
4. Patients with 18.5kg/m^2≤BMI≤40kg/m^2 at the screening visit
5. Patients who have signed an informed consent themselves after receiving detailed explanation about the clinical study

Exclusion Criteria:

1. Patients with type 1 diabetes, secondary diabetes, gestational diabetes, diabetic coma or -pre-coma, metabolic acidosis including lactic acidosis and diabetic ketoacidosis
2. Patients with a medical history of New York Heart Association(NYHA) class III~IV heart failure or with congestive heart failure, acute and unstable heart failure
3. Patients with severe infectious disease or severe traumatic systemic disorders
4. Patients with hypopituitarism or adrenal insufficiency, pulmonary infarction, severe pulmonary dysfunction and other hypoxemia
5. Patients with galactose intolerance, lapp lactase deficiency, glucose-galactose malabsorption
6. Patients with moderate to severe stage renal disease, end stage renal disease, dialysis at the time of screening visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in HbA1c (%) after 24 weeks | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from the baseline in fasting plasma glucose(mg/dL) after 24 weeks | Baseline, 24 weeks
Change from the baseline in HbA1c response rate(<7.0%, <6.5%) after 24 weeks | Baseline, 24 weeks
Change from the baseline in weight after 24 weeks | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si, South Korea